CLINICAL TRIAL: NCT05813106
Title: Effect of Fixed Dose Intravenous Dexmedetomidine on Emergence Delirium After General Anesthesia for a Surgery in Pediatric Patient
Brief Title: Intravenous Dexmedetomidine for Emergence Delirium in Pediatric Patient
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Security Forces Hospital (Other)
Responsible Party: Principal Investigator, Anwar ul Huda, Doctor, Security Forces Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SFH-Dex Peds
Record Dates: First submitted 2023-02-21; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Emergence Delirium; Dexmeditomidine
Keywords: emergence delirium, dexmeditomidine, pediatric patients
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: 2 groups One group will receive IV dexmedetomidine Other control group receive normal saline
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): These patients will receive 0.2 mcg/kg dexmedetomidine intravenously 30 minutes before end
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Control group (Placebo Comparator): These patients will receive normal saline intravenously 30 minutes before end
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Intravenous dexmedetomidine 0.2 mcg/kg
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: normal saline — normal saline
  Arms: Control group

SUMMARY:
Various pharmacological interventions in peri-operative period have been used in literature to prevent ED which include use of propofol, fentanyl, ketamine, clonidine, midazolam and dexmedetomidine etc (5). Dexmedetomidine is a potent highly selective alpha-2 agonist. Its effect on the receptors in brain results in sedation resembling non-REM sleep with minimal respiratory depression (6). It has been used as continuous infusion or as fixed dose in the range between 0.15 mcg/kg to 2 mcg/kg to prevent ED in children (7, 8, 9). Higher doses result in better prevention of ED at the expense of more hemodynamic disturbances and longer PACU stay (9) while lower doses were not as effective (7). The aim of this study was to investigate the role of fixed dose of 0.2 mcg/kg dexmedetomidine in prevention of emergence delirium in pediatric patients undergoing general anesthesia.

DETAILED DESCRIPTION:
Emergence delirium (ED) is an altered state of consciousness that usually occurs within 45 minutes after cessation of anesthesia. It typically presents as disorientation, averted eyes or staring, psychomotor agitation and non-purposeful, resistive movements like pulling, kicking or flailing (1, 2). ED can result in potential risk of bodily harm to patient or healthcare staffs, prolonged PACU (post-anesthesia care unit) stay and postoperative maladaptive changes including temper tantrums, attention seeking, sleep alterations and bed wetting in children (2).

Risk factors for ED include preoperative anxiety and confusion, psychological immaturity and use of various medications peri-operatively (2, 3). The incidence of ED varies by age of patient, anesthesia technique, type of surgeries, pain and also by choice of tool to diagnose ED. It occurs two to three more commonly in children as compared to adults. Scientific literature suggest the incidence of ED in the range between 20 -80 % in pediatric anesthesia practice (4).

Various pharmacological interventions in peri-operative period have been used in literature to prevent ED which include use of propofol, fentanyl, ketamine, clonidine, midazolam and dexmedetomidine etc (5). Dexmedetomidine is a potent highly selective alpha-2 agonist. Its effect on the receptors in brain results in sedation resembling non-REM sleep with minimal respiratory depression (6). It has been used as continuous infusion or as fixed dose in the range between 0.15 mcg/kg to 2 mcg/kg to prevent ED in children (7, 8, 9). Higher doses result in better prevention of ED at the expense of more hemodynamic disturbances and longer PACU stay (9) while lower doses were not as effective (7). The aim of this study was to investigate the role of fixed dose of 0.2 mcg/kg dexmedetomidine in prevention of emergence delirium in pediatric patients undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 2 and 12 years, scheduled to undergo general anesthesia for a surgery with an ASA score of 1 to 3 will be included in the study.

Exclusion Criteria:

* Parents who refused enrollment or later requested removal for the study, those who are unable to give informed consent and patients with known allergy to dexmedetomidine, psychiatric disorders or use of psychiatric medications will not be included in the study

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Emergence delirium | up to 120 minutes
  Emergence delirium will be measured using PAED score

SECONDARY OUTCOMES:
Pain score | every 15 minutes upto discharge from PACU maximum 120 minutes
  VAS pain score
Opioid consumption | upto discharge from PACU maximum 120 minutes
  Morphine equivalent opioid consumption
Side effects | PACU stay maximum 120 minutes
  Side effects including PONV, drowsiness

CONTACTS AND LOCATIONS:
Overall Officials: Anwar ul Huda, FRCA, Principal Investigator — Security Forces Hospital
Locations (1):
- Security Forces Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
We can share IPD on request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication for 6 months
Access Criteria: Direct communication to PI